CLINICAL TRIAL: NCT02367170
Title: Study: Persistent Inflammation, Immunosuppression and Catabolism Syndrome (PICS): A New Horizon for Surgical Critical Care: Project 4A: Inspiratory Muscle Training and Diaphragm Strength
Brief Title: Project 4A: Inspiratory Muscle Training and Diaphragm Strength
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Unable to recruit sufficient number of patients
Sponsor: University of Florida (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB201400889-N; GM111152 (Other Grant/Funding Number: National Institute of General Medical Sciences (NIGMS))
Record Dates: First submitted 2015-01-21; First posted 2015-02-20 (Estimated); Results first posted 2017-01-26 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-04

CONDITIONS: Sepsis
Keywords: respiratory dysfunction; chronic critical illness; diaphragm weakness; sepsis; ventilator dependance
MeSH Terms: conditions — Sepsis; Dyspnea | interventions — Midazolam; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMST Intervention group (Experimental): IMST will be conducted 5 days per week by study staff using a threshold inspiratory muscle training device (Respironics model 735). Prior to training, the tracheal cuff pressure is assessed to ensure no air leakage and appropriate inflation. The IMST training takes approximately 15 minutes to complete. To perform IMST, FiO2 is increased for 2 minutes prior to each training bout to maintain oxygen saturation more than 92%.
  Interventions: Procedure: Bilateral phrenic nerve stimulation and measurement of transdiaphragmatic pressure; Drug: Midazolam; Procedure: Volitional Measurement of Maximal Inspiratory Pressure (MIP); Device: Inspiratory Muscle Strength Training (IMST); Procedure: Diaphragm thickness measurement; Other: Blood and Urine samples
- SHAM group (Sham Comparator): SHAM training will also be conducted five days per week with an identical training device that has been modified by removing the valve leaflet, which essentially removes all inspiratory loading by the device. The modified SHAM device makes a whistling sound during inspiration, which enhances the sham effect. For SHAM treatment, supplemental oxygen FiO2 will be increased for two minute prior to each bout.
  Interventions: Procedure: Bilateral phrenic nerve stimulation and measurement of transdiaphragmatic pressure; Drug: Midazolam; Procedure: Volitional Measurement of Maximal Inspiratory Pressure (MIP); Device: SHAM Inspiratory Muscle Strength Training (IMST); Procedure: Diaphragm thickness measurement; Other: Blood and Urine samples

INTERVENTIONS:
Procedure: Bilateral phrenic nerve stimulation and measurement of transdiaphragmatic pressure — Pressure changes are recorded. The phrenic nerves are stimulated with bilateral magnetic stimulators over the neck. Measurements will be performed on day 1, every 7 days after and on last day of participation. The FiO2 will be increased (at least 20%) for at least 2 min. prior to measurement to maintain oxygen saturation >92%. Prior to activating the stimulator, the artificial airway will be occluded with a pneumatic valve to create a quasi-isometric diaphragm contraction. The airway will be occluded for 3 seconds or less for each stimulation. The procedure will be repeated up to a maximum of 5 times per testing day.
Drug: Midazolam — In the event a subject shows signs of distress during the Bilateral phrenic nerve stimulation and measurement of transdiaphragmatic pressures, a dose of Midazolam is available. IV (in the vein) dose from 0.5 mg to 2 mg.
  Other Names: Versed
Procedure: Volitional Measurement of Maximal Inspiratory Pressure (MIP) — MIP is tested on all subjects on day 1, every 7 days after and on the last day of participation. To measure MIP, a subject will be suctioned, disconnected from the ventilator, and instructed to take a few spontaneous breaths. A 1-way exhalation valve connected to a NICO respiratory monitor will be placed on the ET/tracheotomy tube. The subject will be instructed to inhale and exhale as forcefully as possible for 20 seconds, followed by at least 2 minutes of rest on full mechanical ventilation support. MIP trials will be repeated 3 times, and the greatest negative pressure recorded with a NICO respiratory monitor connected to a laptop computer, which will digitize airway pressure, flow and volume signals at 100Hz. This allows for analysis of the individual pressure waves, facilitating pre-post comparisons of MIP at specific time points during inspiration.
Device: Inspiratory Muscle Strength Training (IMST) — Occurs 5 days/wk using threshold IMST device-Respironics model 735. Prior to training, cuff pressure is assessed, FiO2 increased for 2 min. to keep O2 sats ≥92%. The ventilator circuit is disconnected, IMST device is attached to endotracheal or tracheotomy tube and subject is instructed to exhale then forcefully inhale for 10 breaths. The initial setting of device is set to -5cmH2O, subject must generate a negative inspiratory pressure more negative than -5cmH2O to open spring-loaded valve and receive inspiratory airflow. Pressure setting is made more negative/difficult to open by 2-5cm every few breaths until a setting is found where the patient has difficulty fully opening valve, resulting in valve flutter noise. Training pressure is then made more positive /easier by 2-4cm of H2O, so subject can fully open valve, and 4 sets of 6-10 breaths are completed. Training pressures advanced as rapidly as possible, provided the patient is able to open the valve without"valve flutter"noise.
  Arms: IMST Intervention group
Device: SHAM Inspiratory Muscle Strength Training (IMST) — Training will also be conducted 5 days/wk with an identical IMST device that has been modified by removing the valve leaflet, which essentially removes all inspiratory loading by the device. The modified SHAM IMST device makes a whistling sound during inspiration, which enhances the sham effect. For SHAM treatment, supplemental oxygen FiO2 will be increased for two minute prior to each bout. The ventilator will be disconnected and a SHAM device will be attached to the endotracheal or tracheostomy tube. The subject will be instructed to take 6-10 breaths with a normal tidal volume through the SHAM device and will be reconnected to the ventilator for a 2-minute rest period. The process will be repeated 3 more times for a total of 4 sets of 6-10 breaths.
  Arms: SHAM group
Procedure: Diaphragm thickness measurement — Ultrasound will be used to obtain measurements of the thickness of the right hemidiaphragm. Ultrasonography of the diaphragm will be performed upon enrollment, every 2-4 days during hospitalization and as long as the patient is hospitalized or up to 28 days of participation.
Other: Blood and Urine samples — Peripheral blood and urine samples will be collected once upon study entry day (+/- 2 days), once every 2-4 days and once on final day of study participation (+/- 2days).

SUMMARY:
Investigators will assess the effect of exercise on markers of inflammation and protein catabolism. This research study will further our understanding of how treating Chronic Critical illness (CCI) - related respiratory muscle weakness with strength training can not only improve muscle function, but also potentially blunt the inflammation and catabolism of Peristent Inflammation/Immunosuppression and Catabolism (PICS).

DETAILED DESCRIPTION:
In this research study, investigators will assign study participants to two groups: high intensity inspiratory muscle training and low intensity inspiratory muscle training group. This research study will last up to 28 days in 24 mechanically ventilated patients with CCI. The goal is to determine if the research participants can respond to a training program by improving weaning outcomes from the ventilator. This will be determined by measurement of breathing muscle strength with magnetic stimulation, measurement of diaphragm thickness with ultrasound, inspiratory muscle training, and blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* presence in the surgical or trauma ICU
* age of ≥18 years
* received mechanical ventilation (MV) for 3 days and expected to survive ICU stay
* ability to obtain informed consent from patient or proxy

Exclusion Criteria:

* Inability to speak and understand English
* Uncontrollable source of sepsis with imminent death (e.g., irreversible disease state, unresectable dead bowel)
* Receiving "comfort care only" or have advanced care directives limiting resuscitative efforts
* Known HIV infection with CD4 count < 200 cells/mm
* Organ transplant recipients on immunosuppressive agent(s),
* Known pregnancy
* Unable to follow simple, one-step commands, such as "breathe in as hard as you can!"
* Prior arrangements to be transferred to other facilities before 28 days of treatment
* Contraindications to being disconnected from MV for sham or inspiratory muscle strength training treatment
* Unstable or "difficult airway" at 3 days of ICU care defined by ICU protocol, predicted to last for more than 72 hours
* Ongoing use of vasopressor or vasodilatatory agents for unstable blood pressure. (beyond minimal intermittent amount or "renal perfusion dose,"
* Severe cardiac dysrhythmias
* Esophageal varices or recent esophageal or gastric surgery,
* Upper-airway issues that would be aggravated by inserting esophageal pressure transducers
* Unstable neck/cervical anatomy that might be adversely impacted by bilateral magnetic stimulation of phrenic nerves at the neck
* Acute coronary syndrome
* Pulmonary contraindications (pneumon/hemothorax not drained, flail chest)
* Cardiac pacemakers and/or implanted defibrillator or other implanted electronic devices interfering with magnetic stimulation
* Implanted metal in the chest, neck or head, making magnetic stimulation contraindicated (dental fillings are permitted)
* Postoperative severe surgical problems interfering with the respiratory training (serious postoperative bleeding, wound dehiscence, etc.) - when and if these problems resolve and the patient meets other entry criteria, they will be eligible to be recruited for participation
* Active neuromuscular diseases that would prevent or interfere with responding to strength training (e.g. amyotrophic lateral sclerosis, multiple sclerosis, myasthenia gravis, polymyositis, muscular dystrophy or other dystrophies and myopathies)
* Any other factor that in the investigators' opinions would prevent response to training or create an unsafe condition for the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Martin, Ph.D., PT, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Hospital at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IMST Intervention Group | SHAM Group
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IMST Intervention Group | SHAM Group | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: A Change in Diaphragm Strength From Baseline as an Effect of Inspiratory Muscle Strength Training (IMST) Intervention and Sham Patients
Description: In this randomized, interventional study, 24 CCI patients will be assigned to either a sham group or to receive IMST for up to 28 days. Evaluation of diaphragm/inspiratory muscle strength and muscle thickness will be made with three techniques: 1) non-volitional magnetic stimulation of the phrenic nerves, 2) noninvasive measurement of diaphragm thickness with ultrasound and 3) the standard, clinical method of measuring maximal inspiratory pressure (MIP). Investigators hypothesize that IMST will lead to improvements in all three measures. This study will provide information about possible effective respiratory muscle rehabilitation techniques that are likely to lead to reduced time patients will require mechanical ventilation and improved MIP and weaning outcome in long-term, failure to wean patients
Time Frame: Day 1, Day 3, Day 5, Day 7, Day 9, Day 11, Day 13, Day 14, Day 15, Day 17, Day 19, Day 21, Day 23, Day 25, Day 28
Population: Unable to recruit sufficient number of patients.
Arm/Group | IMST Intervention Group | SHAM Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: A Change in the Results of the Biomarkers of Inflammation From Baseline
Description: Investigators will determine the effects of IMST on biomarkers of inflammation in patients with CCI. Investigators hypothesize that exercise will decrease markers of inflammation compared to the SHAM condition.
Time Frame: Day 1, Day 3, Day 5, Day 7, Day 9, Day 11, Day 13, Day 15, Day 17, Day 19, Day 21
Arm/Group | IMST Intervention Group | SHAM Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: A Change in the Urinary Excretion Markers of Muscle Catabolism From Baseline
Description: Investigators will determine the effects of IMST on urinary excretion markers of muscle catabolism in patients with CCI. Investigators hypothesize that exercise will decrease urinary markers of catabolism compared to the SHAM condition.
Time Frame: Day 1, Day 3, Day 5, Day 7, Day 9, Day 11, Day 13, Day 15, Day 17, Day 19, Day 21
Arm/Group | IMST Intervention Group | SHAM Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | IMST Intervention Group | SHAM Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMST Intervention Group (N=1) | SHAM Group (N=0)
Transitory hypotension (Cardiac disorders) | 1 (1) | 0 (0) — Procedure interrupted to correct hypotension. Subject stabilized and procedure restarted and completed successfully

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No